CLINICAL TRIAL: NCT05044611
Title: AMIloride for the Treatment of Nephrogenic Diabetes Insipidus for Patients With Bipolar Disorder Treated With Lithium: a Randomized Controlled Trial
Brief Title: AMIloride for the Treatment of Nephrogenic Diabetes Insipidus for Patients With Bipolar Disorder Treated With Lithium
Acronym: AMIND
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200042
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Disorder
Keywords: lithium; urine concentration defect
MeSH Terms: conditions — Bipolar Disorder | interventions — Amiloride

STUDY DESIGN:
Intervention Model Description: Two-phased study:
  1st phase: Double blind, placebo-controlled, randomized trial to demonstrate the efficacy of 2 months treatment with amiloride 5mg twice a day to increase urine osmolality in patients with BD treated with lithium for at least 5 years and with a urine concentration defect.
  This double-blinded phase is followed by an open label phase (2nd phase) during 10 months to evaluate the long-term safety profile of the investigated drug and its potential nephroprotective role.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amiloride (Experimental): the experimental arm will receive 5mg of amiloride twice daily during 2 months
  Interventions: Drug: Anhydrous Amiloride Hydrochloride
- Placebo (Placebo Comparator): the control arm will receive a placebo twice daily during 2 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anhydrous Amiloride Hydrochloride — Amiloride is a blocker of ENaC that is administered patients with various disorders, such as primary or secondary hyperaldosteronism. It does not have the market authorization in the indication of lithium-induced NDI.
  Dose : 5 mg Pharmaceutical form: Tablets Daily Posology : 10 mg Route of administration : oral Procedures and duration of treatment: 2 months during the double blinded phase and 10 additional months for the open label phase
  Arms: Amiloride
Drug: Placebo — Route of administration : oral the control arm will receive a placebo twice daily during 2 months
  Arms: Placebo

SUMMARY:
Lithium (Li) is the leading treatment for BD, protecting against both maniac and depressive relapse, and reducing the risk of suicide and mortality. However, despite this major clinical efficacy, the use of lithium is limited by its narrow therapeutic index and by its side effects. Li induces a vasopressin-resistant urinary concentration defect, with resulting nephrogenic diabetes insipidus (NDI) in 12-50 % of patients. This feature is more frequent after 5 years of treatment with lithium. Polyuria and subsequent thirst might affect patients' quality of life, but also cause potentially life-threatening hypernatremia if free access to water is impaired. Thus, we aim at evaluating the efficacy of amiloride on urine concentrating ability in patients with nephrogenic diabetes insipidus due to chronic lithium treatment.

DETAILED DESCRIPTION:
Patients will be referred to the nephrology or the renal physiology department for the usual follow-up of the lithium treatment. After verification of eligilibity criteria, information and collection of consent, patient will be randomized.

During the first phase, patients will be randomized in two parallel groups: the experimental arm will receive 5mg of amiloride twice daily during 2 months and the control arm will receive a placebo twice daily during 2 months.

Measures of fasting urine osmolality will be performed at baseline, 2 months, at 6 months and at 12 months, in order to compare the difference of urine osmolality before and after treatment between the two-randomization arms. Other baseline explorations are as follows: mean number of nocturnal voids, SF-36 questionnaire, thirst intensity and distress scales, YMRS/MADRS mood scale, GAD7 anxiety scale, PSQI sleep scale, GFR measurement and estimation, 24h urine for the quantification of the polyuria and osmolality, plasma and erythrocyte lithium level, serum osmolality, natremia, kaliemia, urea, chlore level, complete blood count, plasma copeptine and vasopressin.

A nephrologist visit will take place 15 days after the initiation of the treatment along with a new measure of plasma lithium level.

Patients will be evaluated at 1 month only if a change in posology is required after the first measurement at day 15 and then at 2, 6 and 12 months.

In parallel, patients will be evaluated by at the psychiatry clinic at 1 month, 2, 6 and 12 months, and in any condition requiring additional visit as usual in standard care (follow-up of anxiety, sleepiness, suicidal ideation, depression).

After the completion of this first phase, the open label second phase will begin. Unblinding the trial will allow the treatment allocation being available for the participants and health care professionals. Amiloride will be continued in participants in the experimental group, and the remaining participants will be followed-up without treatment. This phase will last for 10 months (total trial duration: 12 months).

At one year, renal functions (GFR, urine concentration and 24h urine production) will be assessed along with report of events including hospital admission.

The safety of the experimental treatment will be assessed by regular evaluations of plasma lithium and potassium level, beginning at 2 weeks after treatment initiation and after 2 months. The main risk of amiloride is hyperkalemia, which occurs in patients with severe renal insufficiency. These patients will not be included in our study. Otherwise, the treatment is generally safe and well-tolerated. Plasma lithium level will be measured at the first month clinical evaluation if a change in posology is required after the first measurement at day 15.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 70 years (age ≥ 18 years and <70 years)
* Patient with bipolar disorder
* Patient treated with lithium for at least 5 years
* Patient with a urine concentration defect defined by a maximal urine osmolality < 600 mOsm/kg
* Woman of childbearing age agreeing to use an efficient contraceptive method for 12 months

Exclusion Criteria:

* Renal failure defined as eGFR < 30 ml/min/1.73m² estimated by the CKD-EPI equation
* Kalemia > 5 mmol/l
* Hypersensitivity or known allergy to amiloride
* Hypersensitivity to lactose
* Known adrenal insufficiency
* Concomitant use of other potassium-sparing treatment (e.g. spironolactone, angiotensin converting enzyme inhibitors (ACE), angiotensin II receptor (AT2R) antagonists, calcineurin inhibitors tacrolimus and ciclosporin)
* Acute ongoing infection (less than 3 days before inclusion)
* Severe heart failure (NYHA > II)
* Rhythm, conduction or repolarisation disorder present on an ECG done within 12 months prior to inclusion
* Acute phase of mood disorder
* Uncontrolled diabetes mellitus or diabetes with hyporeninism hypoaldosteronism
* Potassium supplements
* Use of heparins
* Use of trimethoprim
* Cirrhosis
* Oedemas
* Previous use of amiloride use in the 6 months prior to randomisation)
* Pregnant or breastfeeding women
* Participation in another clinical study involving investigational medicinal product or patient being in the exclusion period at the end of a previous study
* Patient refusal to participate
* Non-affiliation to a social security regimen or CMU
* Patient under State Medical Aid
* Subject deprived of freedom, subject under a legal protective measure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
The main objective of this study is demonstrating the efficacy of amiloride to reduce the urine concentration defect in patients treated by lithium and presenting a nephrogenic diabetes insipidus after 2 months of treatment. | 2 month after randomization
  The primary endpoint is the percentage change in maximal urine osmolality before and after 2 months of treatment

SECONDARY OUTCOMES:
Demonstrate the efficacy of amiloride to reduce nocturia | 2 months after randomization and 12 months after randomization
  Difference in mean number of nocturnal voids
Demonstrate the efficacy of amiloride to reduce the sensation of thirst | 2 months after randomization and 12 months after randomization
  Difference in mean number of nocturnal voids
Demonstrate the efficacy of amiloride to reduce polyuria | 2 months after randomization and 12 months after randomization
  Presence of polyuria (defined as a daily urine output > 3 L/day)
Demonstrate the efficacy of amiloride to increase quality of life | 2 months after randomization and 12 months after randomization
  Difference in Quality-of-life scale score (SF36)
Demonstrate the efficacy of amiloride to reduce the decline of eGFR after one year of treatment | 12 months after randomization
  Difference in eGFR (estimated by the CKD-EPI equation based on standardized serum creatinine measurement) before and after 12 months of treatment
Evaluate the effect of amiloride in mood stability | 2 months after randomization and 12 months after randomization
  Difference in Mood Scale scores YMRS
Evaluate the effect of amiloride in circulating lithium levels stability | 2 months after randomization
  Difference in residual plasma lithium levels before and after the 2 months treatment period
Evaluate the effect of amiloride in mood stability | 12 months after randomization
  Total number of hospital admission for maniac or depressive relapse during 12 months of treatment
Evaluate the effect of amiloride in mood stability | 2 months after randomization and 12 months after randomization
  Difference in Mood Scale MADRS
Evaluate the effect of amiloride in mood stability | 2 months after randomization and 12 months after randomization
  Difference in anxiety scale score (GAD7)
Evaluate the effect of amiloride in mood stability | 2 months after randomization and 12 months after randomization
  Difference in the Pittsburgh sleep score (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: DECHANET Aline, Mrs, Study Chair — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (2):
- France (2):
  - Néphrologie, Hôpital Henri-Mondor, Créteil
  - Physiologie Explorations fonctionnelles multidisciplinaires, Hôpital Bichat, Paris

IPD SHARING:
Plan to Share IPD: Undecided